CLINICAL TRIAL: NCT00826631
Title: How Does 4 Weeks of Increased Fast Food Intake Affect Metabolism?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M158-05
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Hyper-Alimentation; Healthy
Keywords: weight; metabolism; cholesterol; insulin
MeSH Terms: conditions — Body Weight; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Fast food intake, doubling of caloric intake, in combination with sedentary behavior (no exercise)
  Interventions: Procedure: Fast food arm
- 2 (No Intervention): Control group, parallel

INTERVENTIONS:
Procedure: Fast food arm — Doubling of regular caloric intake based on fast food, no exercise allowed
  Arms: 1

SUMMARY:
Objective: To study the effect of fast food-based hyper-alimentation on liver enzymes and hepatic triglyceride content (HTGC)and metabolism.

Design: Prospective interventional study with parallel control group. Setting University Hospital of Linköping, Sweden. Participants: 12 healthy men and six healthy women with a mean (SD) age of 26 (6.6) years and a matched control group.

Intervention: Subjects in the intervention group aimed for a body weight increase of 5-15% by eating at least two fast food-based meals a day with the goal to double the regular caloric intake in combination with adoption of a sedentary lifestyle for four weeks.

Main outcome measures: Weekly changes of serum aminotransferases and HTGC measured by proton nuclear magnetic resonance-spectroscopy at baseline and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-obese subjects

Exclusion Criteria:

* General diseases, obesity.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
weight gain | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Linkoping, Linköping, Sweden

REFERENCES:
- [Result] Kechagias S, Ernersson A, Dahlqvist O, Lundberg P, Lindstrom T, Nystrom FH; Fast Food Study Group. Fast-food-based hyper-alimentation can induce rapid and profound elevation of serum alanine aminotransferase in healthy subjects. Gut. 2008 May;57(5):649-54. doi: 10.1136/gut.2007.131797. Epub 2008 Feb 14. PMID 18276725
- [Derived] Lindstrom T, Kechagias S, Carlsson M, Nystrom FH; Fast Food Study Group. Transient increase in HDL-cholesterol during weight gain by hyperalimentation in healthy subjects. Obesity (Silver Spring). 2011 Apr;19(4):812-7. doi: 10.1038/oby.2010.190. Epub 2010 Sep 2. PMID 20814413